CLINICAL TRIAL: NCT06025643
Title: Effects of Electrical Nervous Stimulation Transcutaneous Analysis on Blood Pressure of Patients Hypertensive: Randomized Clinical Trial
Brief Title: Effects of Electrical Nervous Stimulation Transcutaneous in Hypertensive Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other); Leonhardt Ventures LLC (Industry)
Responsible Party: Principal Investigator, Jociane Schardong, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PressureStim
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Hypertension; Hypertension,Essential
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cervical stimulation group (Experimental): TENS will be applied for 30 minutes with a frequency of 5 Hz, pulse width of 200 µs and sufficient intensity to reach the sensory threshold. Ten sessions will be performed over four weeks.
  Interventions: Other: TENS - Cervical stimulation group
- Plus cervical stimulation group (Experimental): TENS will be applied for 30 minutes with a frequency of 5 Hz, pulse width of 200 µs and sufficient intensity to reach the sensory threshold. Ten sessions will be performed over four weeks.
  Interventions: Other: TENS - Plus cervical stimulation group
- Renal stimulation group (Experimental): TENS will be applied for 30 minutes with a frequency of 5 Hz, pulse width of 200 µs and sufficient intensity to reach the sensory threshold. Ten sessions will be performed over four weeks.
  Interventions: Other: TENS - Renal stimulation group
- Control group (No Intervention): This group will not receive any treatment with electrical stimulation.

INTERVENTIONS:
Other: TENS - Cervical stimulation group — TENS will be applied bilaterally through self-adhesive electrodes in the cervicothoracic ganglionic region, located between the C7 and T4 vertebral processes.
  Arms: Cervical stimulation group
Other: TENS - Plus cervical stimulation group — TENS will be applied bilaterally in the cervicothoracic ganglionic region, located between the C7 and T4 vertebral processes, on the earlobe, on the wrists and ankles simultaneously.
  Arms: Plus cervical stimulation group
Other: TENS - Renal stimulation group — TENS will be applied through self-adhesive electrodes in the abdomen (anatomical region corresponding to the kidneys) and dorsal region at the level of the 10th thoracic vertebra.
  Arms: Renal stimulation group

SUMMARY:
Systemic arterial hypertension is a disease characterized by high blood pressure levels. It has a high prevalence, is a precursor of cardiovascular diseases, resulting in high costs to the health system and increased mortality. Transcutaneous electrical nerve stimulation (TENS) is a low-frequency pulsed electrical current widely used for analgesia. Recently, it has been proposed as a non-pharmacological strategy for blood pressure control. The aim of this study is to verify the effect of low-frequency TENS when applied in different anatomical sites on blood pressure, autonomic control and endothelial function in hypertensive patients.

DETAILED DESCRIPTION:
Systemic arterial hypertension is a disease characterized by high blood pressure levels. It has a high prevalence, is a precursor of cardiovascular diseases, resulting in high costs to the health system and increased mortality. Transcutaneous electrical nerve stimulation (TENS) is a low-frequency pulsed electrical current widely used for analgesia. Recently, it has been proposed as a non-pharmacological strategy for blood pressure control. The aim of this study is to verify the effect of low-frequency TENS when applied in different anatomical sites on blood pressure, autonomic control and endothelial function in hypertensive patients. For this, patients will be randomized into 4 groups: group 1 (cervical stimulation), group 2 (plus cervical stimulation ), group 3 (renal stimulation), group 4 (control). Group 1 will receive TENS in the cervical paravertebral region; group 2 will receive stimulation in the cervical paravertebral region, ear lobe, wrist and ankle. Group 3 will have the anatomical region of the kidneys stimulated. Group 4 will not receive any intervention. All the treated patients will receive 30 minutes of stimulation per session, regardless of group allocation. Ten applications will be carried out over the course of a month.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of systemic arterial hypertension: systolic blood pressure (SBP) ≥ 130 mmHg and diastolic blood pressure (DBP) ≥ 80 mmHg diagnosed by ambulatory blood pressure monitoring (ABPM).

Exclusion Criteria:

* Congestive heart failure
* Patients with a cardiac pacemaker
* Previous heart surgery
* Patients with serum creatinine >2.5 mg/dL
* Change in drug therapy in the two months prior to starting the study
* Active smoking

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-10 (Estimated); Primary Completion 2024-02-10 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | Baseline and after 4 weeks
  Systolic blood pressure assessed by ambulatory blood pressure monitoring (ABPM)
Diastolic blood pressure | Baseline and after 4 weeks
  Systolic blood pressure assessed by ambulatory blood pressure monitoring (ABPM)

SECONDARY OUTCOMES:
Autonomic control | Baseline and after 4 weeks
  Autonomic control assessed by analysis of heart rate variability by frequency meter

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo DM Plentz, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre

IPD SHARING:
Plan to Share IPD: No